CLINICAL TRIAL: NCT03505073
Title: Association Between Dietary Habits and Risk Factors for Atherosclerotic Cardiovascular Diseases in Assiut Governorate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Sabry, Assiut - Egypt, Assiut University
Other Study IDs: 10256
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: ASCVD
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Studying and investigating the association between dietary habits and risk factors for atherosclerotic cardiovascular diseases in Assiut governorate

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular diseases (ASCVD) has become the largest single cause of death worldwide. It is responsible for an estimated 17 million deaths and led to 151 million disability-adjusted life years (DALYs) lost (~30.0% of all deaths and 14.0% of all DALYs lost).1 Further, by 2020, 32.0% of the world population deaths will be caused by ASCVD and by 2030; it's expected to be responsible for 33.0% of all deaths (24.2 million).2 Most of atherosclerotic cardiovascular disease events nowadays are taking place in low- and middle-income countries with 80% of the burden occurring in these countries.3

In Egypt, since 1990, ASCVD related mortality was increased over three folds; to be responsible for over 40% of deaths compared with 12% reported two decades earlier.4 Egypt was categorized as a "very-high-risk country for ASCVD" (according to 2016 ESC Guidelines on cardiovascular disease prevention in clinical practice).5 According to (WHO 2014), ASCVD related mortality in Egypt has been increased to account for 46% of total deaths.

Multiple risk factors are attributed to causing ASCVD. These risk factors fall into the categories of either nonmodifiable or modifiable risk factors.6 Nonmodifiable risk factors consist of those conditions that a person cannot alter, including age, heredity, ethnicity and type 1 diabetes.

Whereas modifiable risk factors are conditions that can be altered by making certain lifestyle changes.

In 2003, the Canadian Heart and Stroke Foundation identified nine major modifiable risk factors for ASCVD, namely, tobacco smoking, alcohol abuse, physical inactivity, unhealthy dietary habits, obesity, high BP, high concentrations of dietary fat and blood lipids, and high blood glucose concentrations.7 Sudden stress, frequent migraine and the use of oral contraceptives have also been identified as risk factors for the increased incidence of coronary disease and stroke.8,9 The Egyptian National Hypertension Project (NHP)10,11 was conducted between year 1991 and 1993 in six Egyptian governorates to define the prevalence of ASCVD risk factors in adult Egyptians. The project documented an extremely high prevalence and prominent clustering of ASCVD risk factors in adult men and women particularly obesity.

Since that time, and despite the increasing ASCVD related morbidity and mortality in our Egyptian society, as mentioned before, there's no recent studies (up to our knowledge) was conducted to determine the risk factors associated to ASCVD.

This study overall aim is to systematically explore and investigate the association between dietary habits and risk factors for atherosclerotic cardiovascular diseases in Assiut governorate.

ELIGIBILITY:
- Inclusion criteria: Patients: male or female, aged ≥ 18 years and confirmed to have ASCVD, attending on the outpatient clinics or admitted in Inpatients Ward or ICU of Assiut university Heart Hospital and Assiut Health Insurance Hospital during the study period.

- Exclusion criteria: Patients: aged < 18 years and unconscious patients will be excluded from the study group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients meeting the inclusion criteria attending on the outpatient clinics or admitted in Inpatients Ward or ICU of Assiut university Heart Hospital and Assiut Health Insurance Hospital during the study period.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Detecting the association between dietary habits and risk factors for atherosclerotic cardiovascular diseases in Assiut governorate. | 10 months
  The study's overall aim is to systematically explore and investigate the association between dietary habits and risk factors for atherosclerotic cardiovascular diseases in Assiut governorate.

IPD SHARING:
Plan to Share IPD: Undecided